CLINICAL TRIAL: NCT06340698
Title: Joint Forces to Combat HIV: A Randomized Controlled Trial to Improve the Health-related Quality of Life (HRQoL) of HIV-positive Mothers and Children
Brief Title: Boosting the HRQoL Among HIV+ Mothers and Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: City University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Nancy Xiaonan Yu, Associate Professor, City University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GRF-11606221
Record Dates: First submitted 2024-03-24; First posted 2024-04-01 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: HIV; Perinatal HIV Infection

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Resilience intervention (Experimental): Participants (mother-child dyads) will receive two biweekly sessions of dyadic resilience intervention.
  Interventions: Behavioral: Resilience intervention
- Adherence intervention (Experimental): Participants (mother-child dyads) will receive two biweekly sessions of dyadic adherence intervention.
  Interventions: Behavioral: Adherence intervention
- Control (No Intervention): Participants will receive usual medical treatment.

INTERVENTIONS:
Behavioral: Resilience intervention — Contents of the first session include:
  1. Resilience. Know the concept of resilience.
  2. Stigma management. Discuss stigma experience and learn stigma management strategies such as normalizing the disease.
  3. Self-efficacy. Learn ways of improving self-efficacy, such as experience of success and social support.
  Contents of the second session include:
  1. Mother-child interaction skills. Identify speaking styles that have a negative influence on mother-child interactions. Learn effective communication skills.
  2. Acquiring social support. Know people and resources that could provide support when having HIV-related difficulties and mental health problems.
  3. Emotional regulation. Understand the physiological responses to emotions. Know a range of emotional regulation strategies, such as cognitive reappraisal and deep breathing.
  Arms: Resilience intervention
Behavioral: Adherence intervention — Contents of the first session include:
  1. Adherence behavioral skills. Identify barriers to optimal HAART adherence. Know behavioral skills that can deal with these barriers, such as forgetting, afraid of others' questioning and side effects.
  2. Adherence information and motivation. Know how the HIV virus attack human body and the mechanisms of HAART medication. Understand the influence of adherence level on health outcomes.
  Contents of the second session include:
  1. Adherence motivation. Discuss possibilities and hope of future life, intimate relationship and career.
  2. Mother-child interaction skills. Identify speaking styles that have a negative influence on mother-child interactions concerning HAART medication. Learn effective communication skills.
  3. Acquiring social support. Know people and resources that could provide support when having HAART-related difficulties and problems.
  Arms: Adherence intervention

SUMMARY:
The goal of this randomized controlled trial is to test the effectiveness of a resilience intervention and an adherence intervention in improving health-related quality of life (HRQoL) among perinatally infected HIV positive children and their HIV positive mothers in China.

The main questions it aims to answer are:

1. Whether baseline resilience and treatment adherence are associated with the HRQoL;
2. Whether the resilience intervention will improve the mediators associated with intervention sessions, such as positive coping and social support, the proximal outcome of resilience factors, the distal outcome of HRQoL, and dyadic level outcomes such as dyadic coping;
3. Whether the adherence intervention will improve the mediators associated with intervention sessions, such as adherence information and behavioral skills, the proximal outcome of self-reported adherence, the distal outcome of HRQoL, and dyadic level outcomes such as dyadic coping;
4. Whether the enhanced mediators (e.g., positive coping and social support) associated with the resilience-intervention sessions at the end of the intervention will transmit the effect of the resilience intervention on the increases in resilience factors during follow-ups;
5. Whether the improved mediators (e.g., adherence information and behavioral skills) associated with the adherence-intervention sessions at the completion of the intervention will transmit the effect of the adherence intervention on the increases in adherence in follow-ups.

Participating mother-child dyads in the two intervention arms will receive two sessions of dyadic intervention. Researchers will compare the above-described outcomes between participants in the two intervention arms and the control arm (treatment as usual) to see the effectiveness of the interventions.

ELIGIBILITY:
Inclusion Criteria:

1. the child is HIV positive and perinatally infected, and receives HAART;
2. the biological mother of the child is HIV positive and receives HAART;
3. the mother is a primary caregiver of the child.

Exclusion Criteria:

1. cannot complete the assessment due to a low education level or physical constraints;
2. have been diagnosed with another life-threatening disease (e.g., cancer);
3. have experienced a traumatic event (e.g., a severe car accident or bereavement) in the past 12 months.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Change of health-related quality of life (HRQoL) | Baseline, 2 weeks (immediately after the last session of intervention), 1 month and 3 months
  HRQoL will be measured by the Chinese short version of the World Health Organization Quality of Life (Whoqol Group, 1998). Possible scores range from 0 (worst HRQoL) to 104 (Best HRQoL).
Change of depressive symptoms | Baseline, 2 weeks (immediately after the last session of intervention), 1 month and 3 months
  Depressive symptoms will be measured by the Patient Health Questionnaire-9 (Kroenke, Spitzer, & Williams, 2001). Possible scores range from 0 to 27, with a higher score indicating more depressive symptoms.
Change of anxiety symptoms | Baseline, 2 weeks (immediately after the last session of intervention), 1 month and 3 months
  Anxiety symptoms will be measured by the Generalized Anxiety Disorder 7-item version (Spitzer et al., 2006). Possible scores range from 0 to 21, with a higher score indicating more anxiety symptoms.
Change of resilience factors | Baseline, 2 weeks (immediately after the last session of intervention), 1 month and 3 months
  Resilience factors will be measured by the 25-item Connor-Davidson Resilience Scale (Connor & Davidson, 2003). Possible scores range from 0 to 100, with a higher score indicating better resilience.
Change of HAART adherence | Baseline, 2 weeks (immediately after the last session of intervention), 1 month and 3 months
  Adherence will be measured by (a) a visual analog scale asking the level of adherence (Zhang et al., 2020). Possible scores range from 0 (never adhere) to 10 (always adhere); and (b) single-item questions asking about missing and delayed doses in the last three days, seven days (one week) and 30 days (one month). Children will be asked to report their own adherence behaviors, and mothers will be asked to report both their own and their children's.
Change of mediators in the resilience intervention: Perceived stigma | Baseline, 2 weeks (immediately after the last session of intervention)
  Perceived stigma will be assessed by the 8-item HIV Stigma Scale (Berger et al., 2001; Li et al., 2016). Possible scores range from 8 to 32, with a higher score indicating a higher level of perceived stigma.
Change of mediators in the resilience intervention: Emotional regulation | Baseline, 2 weeks (immediately after the last session of intervention)
  Emotional regulation will be assessed by the Emotional Management Strategy Questionnaire (Fabrizio et al., 2015). Possible scores range from 10 (worst emotional regulation) to 60 (best emotional regulation).
Change of mediators in the resilience intervention: Positive coping | Baseline, 2 weeks (immediately after the last session of intervention)
  Positive coping will be assessed by a combination of the positive reappraisal subscale from the Cognitive Emotion Regulation Questionnaire (Garnefski et al., 2002; Zhu et al., 2008) and the Emotional Processing Subscale from the Emotional Approach Coping Scales (Stanon et al., 2000; Tse et al., 2020). Possible scores range from 8 to 40, with a higher score indicating better positive coping.
Change of mediators in the resilience intervention: Social support | Baseline, 2 weeks (immediately after the last session of intervention)
  Social support will be assessed by a combination of the Perceived Social Support Scale (Blumenthal et al., 1987; Huang, Jiang, & Ren, 1996), the possible scores of which range from 0 (lowest level of support) to 72 (highest level of support), and the usage of support subscale of the Social Support Assessment Scale (Xiao & Yang, 1987), the possible scores of which range from 3 (lowest level of support utilization) to 12 (highest level of support utilization)
Change of mediators in the resilience intervention: Self-efficacy | Baseline, 2 weeks (immediately after the last session of intervention)
  Self-efficacy will be assessed by the General Self-Efficacy Scale (Schwarzer & Aristi, 1997). Possible scores range from 10 to 40, with a higher score indicating a higher level of efficacy.
Change of mediators in the adherence intervention: Adherence information, motivation, and behavioral skills | Baseline, 2 weeks (immediately after the last session of intervention)
  Adherence information, motivation, and behavioral skills will be assessed by the LifeWindows Information-Motivation-Behavioral Skills Antiretroviral Therapy Adherence Questionnaire (LifeWindows Project Team, 2006; Peng et al., 2020). Possible scores of the information, motivation, and behavioral skills subscale range from 9 to 45, 8 to 40, and 13 to 65, respectively, with a higher score indicating a higher level of information, motivation, and behavioral skills.
Change of mediators in the adherence intervention: Illness perception | Baseline, 2 weeks (immediately after the last session of intervention)
  Illness perception will be assessed by the Brief Illness Perception Questionnaire (Broadbent et al., 2006). Possible scores of each of the eight items range from 0 to 10, and each item will be used separately.
Change of mediators in the adherence intervention: Adherence efficacy | Baseline, 2 weeks (immediately after the last session of intervention)
  Adherence efficacy will be assessed by the HIV Treatment Adherence Self-Efficacy Scale (Johnson et al., 2007; Sun et al., 2016). Possible scores range from 0 to 120, with a higher score indicating a higher level of perceived efficacy.
Change of mediators in the adherence intervention: Children's medication-taking responsibility | Baseline, 2 weeks (immediately after the last session of intervention)
  Children's medication-taking responsibility perception and allocation (between mother and child) will be assessed by two visual analog scales respectively. Possible scores of each item range from 0 to 10, with a higher score indicating more self-responsibility than mother-responsibility.

SECONDARY OUTCOMES:
Change of mother-child relationship and interaction: Dyadic coping | Baseline, 2 weeks (immediately after the last session of intervention), 1 month and 3 months
  Dyadic coping will be assessed by two subscales from the Dyadic Coping Inventory (Bodenmann, 2008), namely the common dyadic coping and the evaluation of the dyadic coping subscale. Possible scores range from 7 to 35, with a higher score indicating a higher level of dyadic coping.
Change of mother-child relationship and interaction: Mother-child closeness | Baseline, 2 weeks (immediately after the last session of intervention), 1 month and 3 months
  Mother-child closeness will be assessed by the Closeness subscale of the Network of Relationships-Relationship Quality Version (Buhrmester & Furman, 2008; Kong et al., 2012), the possible scores of which range from 15 (lowest level of closeness) to 90 (highest level of closeness) and the Inclusion of Other in the Self Scale (Aron, A., Aron, N., & Smollan, 1992), the possible scores of which range from 1 (lowest level of closeness) to 7 (highest level of closeness).
Change of mother-child relationship and interaction: Family harmony | Baseline, 2 weeks (immediately after the last session of intervention), 1 month and 3 months
  Family harmony will be assessed by the Family Harmony Scale (Kavikondala et al., 2016). Possible scores range from 10 to 60, with a higher score indicating a higher level of harmony.
Change of mother-child relationship and interaction: Mother-child conflict | Baseline, 2 weeks (immediately after the last session of intervention), 1 month and 3 months
  Mother-child conflict will be measured by the frequency and intensity of parent-child conflicts (Yau & Smetana, 1996), the possible scores of which range from 2 (no conflict) to 10 (highest level of conflict).
Change of mother-child relationship and interaction: Relationship satisfaction | Baseline, 2 weeks (immediately after the last session of intervention), 1 month and 3 months
  Relationship satisfaction will be assessed by a single-item relationship ladder. Possible scores range from 0 to 10, with a higher score indicating a higher level of satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaonan N. Yu, Dr., Principal Investigator — City University of Hong Kong
Locations (1):
- Guangxi Center for Disease Prevention and Control, Nanning, Guangxi, China

IPD SHARING:
Plan to Share IPD: No